CLINICAL TRIAL: NCT01836536
Title: Analysis of Different Circulating Immune Cells in Patients With Recurrent Glioblastoma or Mixed Anaplasic Glioma Treated With Bevacizumab and Search for a Link With Response to Treatment
Brief Title: Search for a Link Between Response to Treatment and Circulating Leucocytes in High Grade Glioma Patients
Acronym: AVA-CELL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center Eugene Marquis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AVA-CELL
Record Dates: First submitted 2012-09-12; First posted 2013-04-22 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Glioblastoma; Glioma
Keywords: High grade glioma; Bevacizumab; Chemotherapy; Myeloid Cells; Treg
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BEVACIZUMAB (Other): BEVACIZUMAB standard of care
  Interventions: Drug: Bevacizumab standard of care

INTERVENTIONS:
Drug: Bevacizumab standard of care — Standard treatment associated with circulating leucocytes (blood samplings)
  Other Names: Avastin

SUMMARY:
Bevacizumab, a monoclonal antibody against vascular endothelial growth factor (VEGF), is an antiangiogenic treatment currently proposed to recurrent high grade glioma patients. Unfortunately some patients fail to respond to this treatment and finding biological factors allowing the discrimination between potential responders and non responders would be very helpful. As the immune system plays a key role in angiogenesis induction and maintenance in cancer, it could serve as a surrogate marker of angiogenesis in cancer patients.

The purpose of this study is to determine the influence of bevacizumab treatment on circulating immune cells in high grade glioma patients and to search for a link between the variation of these cells and the response to treatment.

DETAILED DESCRIPTION:
The following leucocyte subsets will be analyzed in whole blood before treatment and before cycles 3, 5 and 7:

* Classical, intermediate, nonclassical and Tie2 expressing monocytes.
* Regulatory T cells (Treg).
* Myeloid Derived Suppressor cells (MDSCs) The variation of the absolute numbers (or relative percentages) of the cells in the blood of patients will be correlated to the response to treatment assessed according to the RANO criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proved recurrent glioblastoma or anaplasic glioma,
* Tumor recurrence documented by MRI at least 3 months after the end of radiotherapy or chemotherapy.
* Patients for whom a treatment by bevacizumab is proposed by a multidisciplinary team staff.
* Age ≥ 18.
* Signed informed consent.
* Affiliation to a social security coverage

Exclusion Criteria:

* Known Hepatitis B or C or HIV.
* Inclusion in another clinical trial.
* Patient having received an anti-angiogenic therapy.
* Pregnant or breast-feeding woman.
* Person deprived of liberty or under guardianship or trusteeship or judicial protection
* Inability to give informed consent
* Person unable or unwilling to comply with the requirements of the protocol for geographical, social or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-09; Primary Completion 2015-03 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
blood cells populations | up to 4 months
  Analysis of blood cells populations variation during treatment with bevacizumab. Last sampling planned before the 7th cycle of bevacizumab.

SECONDARY OUTCOMES:
Cells variation and RMI response | 6 weeks
  Relationship between variation of blood cells and RMI response after 6 weeks of treatment
Survival | Patients will be followed up from the date of randomization up to their death, assessed up to 100 months
  Link between variation of analyzed cellular population and survival.

CONTACTS AND LOCATIONS:
Overall Officials: Veronique QUILLIEN, MD, Principal Investigator — Center Eugene Marquis
Locations (2):
- France (2):
  - Hôpital Avicenne, Bobigny
  - Center Eugene Marquis, Rennes